CLINICAL TRIAL: NCT02839304
Title: A Prospective, Multicenter Investigation of the Adagio Cryoablation System in Patients With Atrial Fibrillation
Brief Title: Investigation of the Adagio Cryoablation System in Patients With Atrial Fibrillation
Acronym: CryoCure2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Adagio Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS-029
Record Dates: First submitted 2016-07-14; First posted 2016-07-20 (Estimated); Last update posted 2021-09-20 (Actual); Status verified 2019-05

CONDITIONS: Atrial Fibrillation; Atrial Flutter
MeSH Terms: conditions — Atrial Fibrillation; Atrial Flutter

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Catheter Ablation Treatment (Experimental): Cryoablation System: Atrial Fibrillation Ablation
  Interventions: Device: Cryoablation System

INTERVENTIONS:
Device: Cryoablation System — Pulmonary Vein Isolation, Posterior Wall Isolation. May Include Mitral Line ablation, AF Driver ablation, and Cavo-tricuspid Isthmus ablation as indicated

SUMMARY:
The objective of the study is to demonstrate the safety and feasibility of the Adagio Cryoablation System is subjects with Paroxysmal (PAF), Persistent (PsAF) and Long-Standing Persistent Atrial Fibrillation.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is diagnosed with paroxysmal (PAF), persistent, or long standing persistent atrial fibrillation (PsAF) for which an ablation procedure was deemed most appropriate therapy. Paroxysmal AF is defined as recurrent atrial fibrillation (AF) that terminates spontaneously within seven (7) days. Persistent AF is defined as: an episode lasting longer than seven (7) days, but less than one (1) year documented by consecutive ECG recordings of 100% AF greater than seven (7) days apart or an episode requiring electrical or pharmacological cardioversion after 48 hours of AF documented by continuous recording. Long-Standing Persistent AF is defined as continuous AF that lasts longer than one (1) year.
2. Reported incidence of at least one (1) documented episode of symptomatic atrial fibrillation (AF) during the twelve months preceding trial entry (should be documented by rhythm strip or ECG).
3. Failure of at least one anti-arrhythmic medication (AAD) for paroxysmal atrial fibrillation [class I or III, or AV nodal blocking agents such as beta blockers (BB) and calcium channel blockers (CCB)] as evidenced by recurrent symptomatic paroxysmal atrial fibrillation, or intolerable side effects due to AAD.
4. Left atrial size <55 mm in largest dimension as measured and image documented by preoperative imaging (CT, MRI and/or TTE)
5. Left Ventricular Ejection Fraction ≥ 40% (obtained within 12 months prior to the procedure).
6. Anticoagulation therapy: patient is receiving anticoagulation therapy four (4) weeks prior to the ablation procedure (where appropriate) according to 2014 AHA/ACC/HRS Guideline for the Management of Patients with Atrial Fibrillation.
7. Patient is at least 18 and ≤80 years of age.
8. Patient is able and willing to comply with mandatory pre and post follow-up testing.
9. Patient is able and willing to give informed consent.

Exclusion Criteria:

1. Patient had any previous left atrial ablation.
2. History of any valvular cardiac surgical procedure, atrial septal defect closure device; or left atrial appendage closure device.
3. Coronary artery bypass grafting (CABG) procedure within the last 3 months.
4. Awaiting cardiac transplantation or other cardiac surgery within the next 12 months.
5. Atrial clot/thrombus on imaging such as on a trans-esophageal echocardiogram (TEE) performed within 48 hours of the procedure if deemed appropriate by the investigator.
6. History of a documented thromboembolic event within the past one (1) year.
7. Diagnosed atrial myxoma.
8. Patient has defibrillator implant.
9. Patient has known cryoglobulinemia.
10. Patient has any contraindication for oral anticoagulation.
11. Anaphylactic allergy to contrast media.
12. Significant pulmonary disease, (e.g. restrictive pulmonary disease, constrictive or chronic obstructive pulmonary disease) or any other disease or malfunction of the lungs or respiratory system that produces chronic symptoms.
13. Significant congenital anomaly or medical problem that in the opinion of the investigator would preclude enrollment in this study.
14. Acute illness or active systemic infection or sepsis.
15. Unstable angina.
16. Myocardial infarction within the previous three months.
17. History of blood clotting or bleeding abnormalities.
18. Uncontrolled heart failure or New York Heart Association (NYHA) class III or IV heart failure.
19. An intracardiac thrombus, tumor, or other abnormality that precludes catheter introduction or manipulation.
20. Presence of a condition that precludes vascular access
21. Patient has renal dysfunction with glomerular filtration rate < 30 ml/min/1.73m2.
22. Structural heart disease of clinical significance including congenital heart disease where either the underlying abnormality or its correction prohibits or increases the risk of ablation.
23. Atrial fibrillation (AF) secondary to electrolyte imbalance, thyroid disease, or reversible or non-cardiac cause (e.g. surgery, pericarditis).
24. Any history of a cerebrovascular disease, including stroke or Transient Ischemic Attack.
25. Patients with chronic obstructive pulmonary disease (COPD).
26. Continued need for Amiodarone therapy post procedure.
27. Women who are pregnant (by history of menstrual period or pregnancy test if the history is considered unreliable).
28. Any anatomical abnormality of the patient's esophagus which might interfere with esophageal warming balloon insertion, positioning or inflation.
29. Enrollment in an investigational study evaluating another device or drug.
30. Life expectancy less than 12 months.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-07; Primary Completion 2020-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
The primary safety endpoint will be determined by evaluating the incidence of procedural adverse events. | 1 day
The primary safety endpoint will be determined by evaluating the incidence of serious adverse events within 7 days of procedure | 7 days
The primary safety endpoint will be determined by evaluating the incidence of serious adverse events > 7 days after the procedure | 30 days
The primary safety endpoint will be determined by evaluating the incidence of serious adverse events > 30 days after the procedure | 12 months
Technical performance assessed by complete electrical isolation of all pulmonary veins (entrance block). | 1 day
Technical performance assessed by AF termination targeting driver regions, when applicable | 1 day
Technical performance assessed by complete linear block of linear lesions if deployed | 1 day

SECONDARY OUTCOMES:
Performance assessed by percentage of RF focal ablation (touch up) to reach the primary performance endpoint. | 1 day
Performance assessed by procedural fluoroscopy times | 1 day
Performance assessed by ablation times | 1 day
Performance assessed by total procedure times) | 1 day
Performance assessed by complete freedom from documented AF or other atrial tachycardia (>30s), using a Holter monitor at 6-, 9-, and 12 months post ablation, after a single procedure and off AAD (following a 3 month blanking period). | 12 months

CONTACTS AND LOCATIONS:
Locations (3):
- OLV Hospital, Aalst, Belgium
- Cardiology Hospital of Haut-Lévêque, Pessac, France
- St. Antonius Hospital, Nieuwegein, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Klaver MN, De Potter TJR, Iliodromitis K, Babkin A, Cabrita D, Fabbricatore D, Boersma LVA. Ultralow temperature cryoablation using near-critical nitrogen for cavotricuspid isthmus-ablation, first-in-human results. J Cardiovasc Electrophysiol. 2021 Aug;32(8):2025-2032. doi: 10.1111/jce.15142. Epub 2021 Jul 9. PMID 34196991